CLINICAL TRIAL: NCT00638183
Title: Special Survey Long-term Treatment
Brief Title: Special Survey Long-term Treatment With Tiotropium on COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.315
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2010-04-05 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Since Spiriva Inhalation Capsules 18mcg (hereinafter this product) are indicated for treatment of patients with chronic obstructive pulmonary disease (i.e. patients with chronic bronchitis or pulmonary emphysema) and usually intended for long-term use, the present survey is conducted to collect safety and effectiveness information on the use of this product for long period of time in daily clinical settings, and to obtain proper drug use information.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Chronic Obstructive Pulmonary Disease
2. Patients were expected to use the product for long period of time

Exclusion Criteria:

1. Patients with glaucoma
2. Patients with micturition disorder due to prostatic hyperplasia etc.
3. Patients with a history of hypersensitivity to atropine or its derivatives or to any component of this product

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COHORT
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (89):
- Japan (89):
  - Boehringer Ingelheim Investigational Site, Asahikawa
  - Boehringer Ingelheim Investigational Site, Chikushino-shi
  - Boehringer Ingelheim Investigational Site, Daitō
  - Boehringer Ingelheim Investigational Site, Ebina
  - Boehringer Ingelheim Investigational Site, Echizen
  - Boehringer Ingelheim Investigational Site, Fukui
  - Boehringer Ingelheim Investigational Site, Fukushima
  - Boehringer Ingelheim Investigational Site, Funabashi
  - Boehringer Ingelheim Investigational Site, Gosen
  - Boehringer Ingelheim Investigational Site, Habikino
  - Boehringer Ingelheim Investigational Site, Hakodate
  - Boehringer Ingelheim Investigational Site, Hayashimacho
  - Boehringer Ingelheim Investigational Site, Higashiosakaka
  - Boehringer Ingelheim Investigational Site, Himeji
  - Boehringer Ingelheim Investigational Site, Hirosaki
  - Boehringer Ingelheim Investigational Site, Hiroshima
  - Boehringer Ingelheim Investigational Site, Hitachi
  - Boehringer Ingelheim Investigational Site, Iizuka
  - Boehringer Ingelheim Investigational Site, Ikoma
  - Boehringer Ingelheim Investigational Site, Ishinomaki
  - Boehringer Ingelheim Investigational Site, Itanocho
  - Boehringer Ingelheim Investigational Site, Kasukabe
  - Boehringer Ingelheim Investigational Site, Katsuragichō
  - Boehringer Ingelheim Investigational Site, Kawasaki
  - Boehringer Ingelheim Investigational Site, Kishiwada
  - Boehringer Ingelheim Investigational Site, Kitakyushu
  - Boehringer Ingelheim Investigational Site, Kobayashi
  - Boehringer Ingelheim Investigational Site, Koga
  - Boehringer Ingelheim Investigational Site, Komaki
  - Boehringer Ingelheim Investigational Site, Komatsu
  - Boehringer Ingelheim Investigational Site, Kōshū
  - Boehringer Ingelheim Investigational Site, Kumamoto
  - Boehringer Ingelheim Investigational Site, Kunimichō
  - Boehringer Ingelheim Investigational Site, Kyoto
  - Boehringer Ingelheim Investigational Site, Kyōtango
  - Boehringer Ingelheim Investigational Site, Matsudo
  - Boehringer Ingelheim Investigational Site, Matsue
  - Boehringer Ingelheim Investigational Site, Matsumoto
  - Boehringer Ingelheim Investigational Site, Mihamacho
  - Boehringer Ingelheim Investigational Site, Minamiuonuma
  - Boehringer Ingelheim Investigational Site, Mishima
  - Boehringer Ingelheim Investigational Site, Mizumakimachi
  - Boehringer Ingelheim Investigational Site, Morioka
  - Boehringer Ingelheim Investigational Site, Nagaoka
  - Boehringer Ingelheim Investigational Site, Nagasaki
  - Boehringer Ingelheim Investigational Site, Nagoya
  - Boehringer Ingelheim Investigational Site, Nichinan
  - Boehringer Ingelheim Investigational Site, Niihama
  - Boehringer Ingelheim Investigational Site, Nōgata
  - Boehringer Ingelheim Investigational Site, Numata
  - Boehringer Ingelheim Investigational Site, Obihiro
  - Boehringer Ingelheim Investigational Site, Odawara
  - Boehringer Ingelheim Investigational Site, Osaka
  - Boehringer Ingelheim Investigational Site, Ōbu
  - Boehringer Ingelheim Investigational Site, Ōgaki
  - Boehringer Ingelheim Investigational Site, Ōkuchi
  - Boehringer Ingelheim Investigational Site, Ōtsu
  - Boehringer Ingelheim Investigational Site, Saiki
  - Boehringer Ingelheim Investigational Site, Saitama
  - Boehringer Ingelheim Investigational Site, Sakai
  - Boehringer Ingelheim Investigational Site, Sakede
  - Boehringer Ingelheim Investigational Site, Sapporo
  - Boehringer Ingelheim Investigational Site, Sayama
  - Boehringer Ingelheim Investigational Site, Sendai
  - Boehringer Ingelheim Investigational Site, Shiroishi
  - Boehringer Ingelheim Investigational Site, Shiroishichō
  - Boehringer Ingelheim Investigational Site, Shizuoka
  - Boehringer Ingelheim Investigational Site, Tagawa
  - Boehringer Ingelheim Investigational Site, Takarazuka
  - Boehringer Ingelheim Investigational Site, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Higashiyamato
  - Boehringer Ingelheim Investigational Site, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Kita-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Koto-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Otaku-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site, Tsu
  - Boehringer Ingelheim Investigational Site, Tsukuba
  - Boehringer Ingelheim Investigational Site, Ube
  - Boehringer Ingelheim Investigational Site, Uji
  - Boehringer Ingelheim Investigational Site, Urayasu
  - Boehringer Ingelheim Investigational Site, Uruma
  - Boehringer Ingelheim Investigational Site, Utsunomiya
  - Boehringer Ingelheim Investigational Site, Yamagata
  - Boehringer Ingelheim Investigational Site, Yame
  - Boehringer Ingelheim Investigational Site, Yokohama
  - Boehringer Ingelheim Investigational Site, Yorocho
  - Boehringer Ingelheim Investigational Site, Yurihonjō

RESULTS

PARTICIPANT FLOW:
Groups:
- Spiriva Treatment: Daily Therapy
Period: Overall Study
Arm/Group | Spiriva Treatment
Started | 385
Completed | 266
Not Completed | 119
Not completed — Adverse Event | 23
Not completed — Lack of Efficacy | 14
Not completed — Physician Decision | 9
Not completed — Lost to Follow-up | 46
Not completed — Other reason not defined above | 27

BASELINE CHARACTERISTICS:
Population: Number of participants in this summary is "Number of patients eligible for efficacy analysis"
  Throughout this report, the discrepancy between the total number of participants and the numbers analyzed for a certain parameter is due to missing data.
Arm/Group | Spiriva Treatment
Number analyzed (Participants) | 249
Age, Customized [Number; unit: Participants]
  <65 years | 51
  65≤ to <75 years | 88
  >=75 years | 103
  Unknown | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 212

OUTCOME MEASURES:

1. Secondary Outcome: Effective Rate of Comprehensive Evaluation
Description: Evaluate from improvement FEV1 (forced expiratory volume in 1 second) and/or Symptoms by Investigator.
  Latest time point, at the end of the observation or 1 year after the initiation of treatment, investigator judged and decided "comprehensive evaluation".
  "comprehensive evaluation" was classified into 3 category, "improve" "No change+Aggravated" and "Unassessable" by reference to the result of FEV1 and symptoms. The effective rate was derived from rate of "Improvement" in total number of analyzed patients
Time Frame: 52 weeks
Population: 249 patient were evaluated the efficacy
Measure: Number; unit: percentage of effective patients
Arm/Group | Spiriva Treatment
Number analyzed (Participants) | 249
percentage of effective patients | 70.9

2. Secondary Outcome: Change in Forced Expiratory Volume (L) in 1 Second at 52 Weeks
Description: Difference between Mean of Pre- and each week's forced expiratory volume in 1 second (FEV1) The FEV1 is the volume (Liters) exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. FEV1 is by far the most frequently used index for assessing airway obstruction, bronchoconstriction or bronchodilatation
Time Frame: Pre treatment and 52 weeks after the treatment
Population: All patients for which respiratory function testing was conducted at baseline and at 52 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Spiriva Treatment
Number analyzed (Participants) | 111
Liters | 0.119 (0.208)

3. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: Number of patients with AEs
Time Frame: Pre treatment and 52 weeks after the treatment
Population: 373 patients were involved in the safety analysis data
Measure: Number; unit: Participants
Arm/Group | Spiriva Treatment
Number analyzed (Participants) | 373
Participants | 71

4. Primary Outcome: Number of Patients With Adverse Drug Reactions (ADRs)
Description: Number of Patients with ADRs. An adverse drug reaction was defined as an adverse event with a relationship to Tiotropium inhalation.
Time Frame: Pre treatment and 52 weeks after the treatment
Population: 373 patients were involved in the safety analysis data
Measure: Number; unit: Participants
Arm/Group | Spiriva Treatment
Number analyzed (Participants) | 373
Participants | 27

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Spiriva Treatment
Serious Adverse Events (participants affected / at risk) | 33/373
Other Adverse Events (participants affected / at risk) | 0/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva Treatment (N=373)
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Macular degeneration (Eye disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Left atrial dilatation (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Death (General disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cor pulmonale (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract